CLINICAL TRIAL: NCT03499158
Title: Role of Terminal Latency Index, Residual Latency and Median Ulnar F Latency Difference in Carpal Tunnel Syndrome
Brief Title: Terminal Latency Index, Residual Latency and Median Ulnar F Latency Difference in Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: ASLIHAN UZUNKULAOGLU (Other)
Collaborators: Baskent University (Other)
Responsible Party: Sponsor-Investigator, ASLIHAN UZUNKULAOGLU, Ufuk University, Ufuk University
Organization: Ufuk University (Other)
Other Study IDs: KA15/280
Record Dates: First submitted 2018-04-11; First posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: affected arms of patients who had gone to electrodiagnostic study and diagnosed as carpal tunnel syndrome
  Interventions: Other: nerve conduction study
- 2: healthy arms of patients who had gone to electrodiagnostic study and diagnosed as carpal tunnel syndrome in the other arms
  Interventions: Other: nerve conduction study

INTERVENTIONS:
Other: nerve conduction study — nerve conduction study

SUMMARY:
Terminal latency index, residual latency and median ulnar F latency difference in carpal tunnel syndrome are specific parameters for the diagnosis

DETAILED DESCRIPTION:
Carpal tunnel syndrome is the most common compression neuropathy. This study was performed to determine the value of terminal latency index, residual latency and median ulnar F latency difference to investigate their sensitivity and specificity in the diagnosis of this syndrome.

We retrospectively determined the 160 patients. We evaluated the nerve conduction studies of patient and healthy arms. We recorded all nerve conduction study values.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had gone to electrodiagnostic study and diagnosed as carpal tunnel syndrome

Exclusion Criteria:

* any history of hereditary polyneuropathies
* acquired polyneuropathies
* surgery or local steroid injections for upper limbs or effect the study
* any history of fracture at the sites of stimulation or recording

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who had gone to electrodiagnostic study and diagnosed as carpal tunnel syndrome
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-02 (Actual)

PRIMARY OUTCOMES:
nerve conduction studies | one month

IPD SHARING:
Plan to Share IPD: No